CLINICAL TRIAL: NCT00947011
Title: The Effect of Dipeptidyl Peptidase-4 Inhibition on GLP-1 Induced Insulin Secretion and Glucose Turnover During Mild Stable Hyperglycemia in Young and Old Normal Volunteers
Brief Title: Dipeptidyl Peptidase-4 Inhibition on Glucagon-like Peptide-1 (GLP-1)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left JHU
Sponsor: Johns Hopkins University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: NA_00018441
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Glucose Homeostasis
Keywords: Healthy volunteers; GLP-1; Januvia; Sitagliptin
MeSH Terms: interventions — Sugars; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Januvia (Active Comparator)
  Interventions: Drug: Januvia

INTERVENTIONS:
Drug: Placebo — 1 tablet 100 mg once a day
  Other Names: Sugar pill
  Arms: Placebo
Drug: Januvia — 1 tablet 100 mg once a day
  Other Names: Sitagliptin
  Arms: Januvia

SUMMARY:
This research is being done to evaluate the effect of glucagon-like peptide-1 (GLP-1, a naturally occurring hormone) on insulin release and to examine whether there is extra insulin release when GLP-1 is not allowed to be rapidly inactivated.

DETAILED DESCRIPTION:
The purpose of the present proposal is to 1) examine the role of dipeptidyl peptidase (DPP-4) inhibition on insulin release during a hyperglycemic clamp while GLP-1 is being infused and, 2) further elucidate the role of the metabolite of GLP-1, that is GLP-1 9-36 amide (GLP-1m). During stable and very reproducible elevated plasma glucose levels the effect of increased active incretin levels with DPP-4 inhibitors should result in increased plasma insulin levels. Therefore the aim of this protocol is to document whether plasma insulin levels are increased following GLP-1 infusion in the presence or absence of DPP-4 inhibitors. Additionally, the investigators have shown that some improvement in glucose homeostasis during GLP-1 administration is due in part to the metabolite of GLP-1, i.e. GLP-1 (9-36) amide (GLP-1m). Therefore, the investigators will also test the role of the latter by infusing GLP-1m when the volunteers are being treated with DPP-4 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Hct level of at least 34% for women and 36% for men
* Women of non-bearing potential and women of childbearing potential using adequate contraception
* Serum creatine level of less than 1.7 mg/dl
* Four groups:

  * Age 21-45 (BMI between 18.50-24.99) & (BMI between 30-35)
  * Age greater than 65 years (BMI between 18.50-24.99) & (BMI between 30-35)

Exclusion Criteria:

* Pregnant and/or lactating females
* Women of childbearing potential not willing to use adequate contraception
* Hct below inclusion criteria
* Serum creatine level greater than 1.8 mg/dl
* Age less than 21 and age between 46-64
* Diabetes mellitus
* BMI less than 18 and BMI greater than 35

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dariush Elahi, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Although 12 participants were enrolled in this study, their assignment to a specific Arm/Group is unknown, as the PI has left the institution and no further data (if any) is available.
Groups:
- All Participants: Januvia: 1 tablet 100 mg once a day
  OR
  Placebo comparator
Period: Overall Study
Arm/Group | All Participants
Started | 12
Completed | 0
Not Completed | 12
Not completed — Study was terminated,PI left institution | 12

BASELINE CHARACTERISTICS:
Population: Although 12 participants were enrolled in this study, their assignment to a specific Arm/Group is unknown, as the PI has left the institution and no further data (if any) is available.
Groups:
- All Particpants: Januvia: 1 tablet 100 mg once a day
  OR
  Placebo: 1 tablet 100 mg once a day
Arm/Group | All Particpants
Number analyzed (Participants) | 12
Age, Customized [Number; unit: participants]
  >=21 and <=75 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Insulin Release Rate and Hepatic Glucose Release
Time Frame: One year
Population: Data was not collected for this outcome measure. The study was terminated. The P.I. left the institution.
Arm/Group | Januvia | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Peripheral Glucose Utilization and Peripheral Glucagon Release
Time Frame: one year
Population: Data was not collected for this outcome measure. The study was terminated. The P.I. left the institution.
Arm/Group | Januvia | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: This study was prematurely terminated because the P.I. left the institution. The time frame for Adverse Event data (if collected) is unknown.
Description: This study was prematurely terminated because the P.I. left the institution. The data for Adverse Events, if collected, is unknown.
Arm/Group | Januvia | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes